CLINICAL TRIAL: NCT00314249
Title: A Phase III Pivotal, Multicenter, Double-blind, Randomized, Placebo-Controlled Monotherapy Study of Milnacipran for the Treatment of Fibromyalgia.
Brief Title: Study of Milnacipran for the Treatment of Fibromyalgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: Cypress Bioscience, Inc. (Industry)
Responsible Party: Robert Palmer, MD, Forest Research Institute, a subsidiary of Forest Laboratories, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MLN-MD-03
Record Dates: First submitted 2006-04-11; First posted 2006-04-13 (Estimated); Results first posted 2009-11-02 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Milnacipran

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator): Placebo, oral administration, twice daily for 12 weeks
  Interventions: Drug: Placebo
- Milnacipran (Experimental): Milnacipran 100mg/day (50mg BID [twice a day])
  Interventions: Drug: Milnacipran 100mg

INTERVENTIONS:
Drug: Placebo — Placebo, oral administration, twice daily for 12 weeks
  Arms: Placebo
Drug: Milnacipran 100mg — Milnacipran 100mg per day (50mg BID [twice a day])
  Arms: Milnacipran

SUMMARY:
The purpose of this study was to demonstrate the efficacy and safety of milnacipran at a dosage of 100 mg/day in the treatment of the fibromyalgia syndrome or the pain associate with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of fibromyalgia defined by 1990 American College of Rheumatology (ACR) Criteria

Exclusion Criteria:

* psychiatric illness,
* depression,
* suicidal risk,
* substance abuse,
* pulmonary dysfunction,
* renal impairment,
* active cardiac disease,
* liver disease,
* autoimmune disease,
* cancer,
* inflammatory bowel disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1025 (Actual)
Dates: Start 2006-04; Primary Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Forest Investigative Site, Tuscaloosa, Alabama
  - Forest Investigative Site, Fresno, California
  - Forest Investigative Site, Pismo Beach, California
  - Forest Investigative Site, Vista, California
  - Forest Investigative Site, St. Petersburg, Florida
  - Forest Investigative Site, Stuart, Florida
  - Forest Investigative Site, Atlanta, Georgia
  - Forest Investigative Site, Springfield, Massachusetts
  - Forest Investigative Site, Worcester, Massachusetts
  - Forest Investigative Site, Omaha, Nebraska
  - Forest Investigative Site, Haddon Heights, New Jersey
  - Forest Investigative Site, Johnson City, New York
  - Forest Investigative Site, Syracuse, New York
  - Forest Investigative Site, Greensboro, North Carolina
  - Forest Investigative Site, Cleveland, Ohio
  - Forest Investigative Site, Columbus, Ohio
  - Forest Investigative Site, Toledo, Ohio
  - Forest Investigative Site, Eugene, Oregon
  - Forest Investigative Site, Mechanicsburg, Pennsylvania
  - Forest Investigative Site, Anderson, South Carolina
  - Forest Investigative Site, Greer, South Carolina
  - Forest Investigative Site, Richardson, Texas
  - Forest Investigative Site, Virginia Beach, Virginia

REFERENCES:
- [Derived] Saxe PA, Arnold LM, Palmer RH, Gendreau RM, Chen W. Short-term (2-week) effects of discontinuing milnacipran in patients with fibromyalgia. Curr Med Res Opin. 2012 May;28(5):815-21. doi: 10.1185/03007995.2012.677418. Epub 2012 Apr 10. PMID 22429066
- [Derived] Arnold LM, Gendreau RM, Palmer RH, Gendreau JF, Wang Y. Efficacy and safety of milnacipran 100 mg/day in patients with fibromyalgia: results of a randomized, double-blind, placebo-controlled trial. Arthritis Rheum. 2010 Sep;62(9):2745-56. doi: 10.1002/art.27559. PMID 20496365

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was from 4/28/06 through 12/27/07 with last patient last visit on 6/30/08 at 65 centers in the US and 3 centers in Canada
Pre-assignment Details: Upon completion of the washout period, a two-week baseline period was completed prior to randomization. Patients were then randomized in a 1:1 ratio to either placebo or milnacipran 100 mg/day (50 mg BID [twice a day])
Groups:
- Placebo: Placebo administered orally BID (twice a day) for 12 weeks of stable dose treatment phase
- Milnacipran: Milnacipran 100 mg per day, administered orally (BID [twice a day]) for 12 weeks of stable dose treatment phase
Period: Overall Study
Arm/Group | Placebo | Milnacipran
Started | 509 | 516
Completed | 357 | 353
Not Completed | 152 | 163
Not completed — Adverse Event | 73 | 94
Not completed — Lack of Efficacy | 33 | 24
Not completed — Withdrawal by Subject | 21 | 28
Not completed — Lost to Follow-up | 15 | 9
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawn for other reasons | 4 | 1
Not completed — Non-Compliant | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Milnacipran | Total
Number analyzed (Participants) | 509 | 516 | 1025
Age Continuous [Mean (Standard Deviation); unit: years] | 48.73 (10.56) | 49.07 (10.79) | 48.90 (10.67)
Age, Customized [Number; unit: participants]
  <=20 years | 2 | 2 | 4
  Between 20 and 60 years | 437 | 429 | 866
  >=60 years | 70 | 85 | 155
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 477 | 500 | 977
  Male | 32 | 16 | 48
Region of Enrollment [Number; unit: participants]
  United States | 463 | 469 | 932
  Canada | 46 | 47 | 93

OUTCOME MEASURES:

1. Secondary Outcome: Time-Weighted Average of Patient Experience Diary (PED) Reported Morning 24-Hour Recall Pain Scores for Weeks 1-12 of the Stable Dose Phase
Description: Time-weighted average (area under the curve [AUC]) of the weekly average Patient Experience Diary (PED)-reported morning recall pain scores for weeks 1 through 12 of the stable dose treatment phase is the area under the Patient Experience Diary (PED)-time curve estimated using the trapezoidal method and normalized by time.
  PED is the Patient Experience Diary, an electronic diary system used for collection of patient self-reported pain data. Outcome measure is assessed using the VAS Pain Intensity Scale from 0-100 millimeters anchored at 0 mm (no pain) to 100 mm (worst possible pain).
Time Frame: Weeks 1 through 12 of the stable dose treatment phase (Visit TX0-TX12)
Population: The analysis was performed based on intent-to-treat population defined as all randomized patients who took at least one dose of double-blind study medication. For all subjects with missing assessments for weeks 1-12 of the stable dose treatment phase, values were imputed using last observation carried forward (LOCF).
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Placebo | Milnacipran
Number analyzed (Participants) | 509 | 516
units on scale | 48.0 (0.83) | 41.2 (0.87)
Statistical Analysis 1: Comparison: Placebo vs Milnacipran; This parameter was analyzed using an ANCOVA model with treatment group and study center as factors and baseline value as a covariate; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = -6.38, 95% CI [-8.56 to -4.19]

2. Secondary Outcome: Time-Weighted Average of Patient Global Impression of Change (PGIC) From Visit TX0-TX12.
Description: Time-weighted average (area under the curve [AUC]) for Patient Global Impression of Change (PGIC) from Visit TX0-TX12 is the area under the PGIC-time curve estimated using the trapezoidal method and normalized by time.
  PGIC is an efficacy assessment on a scale of 1-7 taken at visits TX0-TX12. The wording of the assessment is as follows: "Since the start of the study, overall my fibromyalgia is:" 1=Very Much Improved, 2=Much Improved, 3=Minimally Improved, 4=No Change, 5=Minimally Worse, 6=Much Worse, and 7-Very Much Worse.
Time Frame: Weeks 1-12 (Visit TX0-TX12) of the stable dose treatment phase
Population: The analysis was performed based on intent-to-treat population defined as all randomized patients who took at least one dose of double-blind study medication. For all subjects with missing assessments from weeks 1-12 of the stable dose treatment phase, values were imputed using last observation carried forward (LOCF).
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Placebo | Milnacipran
Number analyzed (Participants) | 486 | 495
units on scale | 3.4 (0.06) | 2.9 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Milnacipran; This parameter was analyzed using an ANOVA model with treatment group and study center as factors; Test type: Superiority or Other; ANOVA; Mean Difference (Net) = -0.53, 95% CI [-0.69 to -0.38]

3. Secondary Outcome: Change From Baseline in the Multi-Dimensional Fatigue Inventory (MFI) Total Score at Visit TX12.
Description: Change from Baseline in the Multi-Dimensional Fatigue Inventory (MFI) total score at TX12. Negative differences indicate decrease of fatigue.
  MFI is a subjective report of fatigue symptoms consisting of 20 items that can be scored to produce 5 dimensions: general fatigue, physical fatigue, mental fatigue, reduced motivation, and reduced activity. The MFI is a 1-5 scale with 1="yes, that is true" and 5="no, that is not true."
Time Frame: Baseline through end of week 12 (Visit TX12)
Population: The analysis was performed based on intent-to-treat population defined as all randomized patients who took at least one dose of double-blind study medication. For all subjects with missing assessments at the end of week 12 (Visit TX12), values were imputed using Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Placebo | Milnacipran
Number analyzed (Participants) | 502 | 508
units on scale | -3.96 (0.549) | -5.50 (0.599)
Statistical Analysis 1: Comparison: Placebo vs Milnacipran; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = -1.69, 95% CI [-3.27 to -0.11]

4. Primary Outcome: Composite Syndrome Responder Status
Description: Composite Syndrome Responder Status is the number of responders based on 3 domains: (1) 30% reduction in pain (as recorded in the Patient Experience Diary [PED], electronic diary, during the morning report; 24 hour recall); (2) patient global impression of change (PGIC) score of "very much improved" and "much improved;" and (3) physical function improvement of 6 or more points on Short Form-36 Physical Component Summary (SF-36 PCS)
Time Frame: At the end of the three-month stable dose treatment phase
Population: The primary efficacy analysis was performed based on intent-to-treat population defined as all randomized patients who took at least one dose of double-blind study medication. All subjects with missing assessments at the end of the three-month stable dose treatment phase were considered non-responders (baseline value carried forward (BOCF)).
Measure: Number; unit: Syndrome Responder Participants
Arm/Group | Placebo | Milnacipran
Number analyzed (Participants) | 509 | 516
Syndrome Responder Participants | 56 | 103
Statistical Analysis 1: Comparison: Placebo vs Milnacipran; The test of no difference in the responder rate between milnacipran and placebo groups was performed using a logistic regression model with treatment group, baseline pain score, and baseline SF-36 PCS score as explanatory variables; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Closed testing procedure used to control overall type 1 error rate at 5%: fibromyalgia syndrome tested prior to fibromyalgia pain; Odds Ratio (OR) = 2.06, 95% CI [1.45 to 2.94]

5. Primary Outcome: Composite Pain Responder Status
Description: Composite Pain Responder Status is the number of responders based on two domains: (1) 30% reduction in pain (as recorded in the Patient Experience Diary [PED], electronic diary, during the morning report; 24 hour recall); and (2) Patient Global Impression of Change (PGIC) score of "very much improved" or "much improved."
Time Frame: At the end of three-month stable dose treatment phase
Population: The primary efficacy analysis was performed based on intent-to-treat population defined as all randomized patients who took at least one dose of double-blind study medication. All subjects with missing assessments at the end of three-month stable dose treatment phase were considered non-responders (baseline value carried forward (BOCF)).
Measure: Number; unit: Pain Responder Participants
Arm/Group | Placebo | Milnacipran
Number analyzed (Participants) | 509 | 516
Pain Responder Participants | 90 | 147
Statistical Analysis 1: Comparison: Placebo vs Milnacipran; The test of no difference in the responder rate between milnacipran and placebo groups was performed using a logistic regression model with the treatment group and baseline pain score as explanatory variables; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Closed testing procedure was used to control overall type 1 error rate at 5%: fibromyalgia pain tested after statistically significant fibromyalgia syndrome test; Odds Ratio (OR) = 1.86, 95% CI [1.38 to 2.51]

6. Secondary Outcome: Time-Weighted Average of the Short Form-36 Physical Component Summary (SF-36 PCS) Score From Visit TX0-TX12
Description: Short Form-36 (SF-36): pt. questionnaire (36 questions) which give rise to 8 domains & 2 component summaries (mental and physical); assessing quality of life, health & functional status.
  SF-36 PCS: weighted summary of physical function using all 8 domains.
  Scores are standardized so that the range for all domains and component summaries is 0 (worst possible score) to 100 (best possible score). Higher scores indicate better health or functional status.
  SF-36 PCS AUC (Area under the Curve): estimated using trapezoidal method, normalized by time.
Time Frame: Weeks 1-12 (Visit TX0-TX12) of the stable dose treatment phase
Population: The analysis was performed based on intent-to-treat population defined as all randomized patients who took at least one dose of double-blind study medication. For all subjects with missing assessments from weeks 1-12 (Visit TX0-TX12) of the stable dose treatment phase, values were imputed using the Last Observation Carried Forward (LOCF) approach.
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Placebo | Milnacipran
Number analyzed (Participants) | 509 | 516
units on scale | 36.4 (0.37) | 37.9 (0.37)
Statistical Analysis 1: Comparison: Placebo vs Milnacipran; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = 1.65, 95% CI [0.86 to 2.44]

ADVERSE EVENTS:
Arm/Group | Placebo | Milnacipran
Serious Adverse Events (participants affected / at risk) | 7/509 | 10/516
Other Adverse Events (participants affected / at risk) | 382/509 | 434/516
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=509) | Milnacipran (N=516)
Anxiety (Psychiatric disorders) | 0 | 1
Apendicitis (Infections and infestations) | 1 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chest Pain (General disorders) | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Confusional State (Psychiatric disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Embolic Cerebral Infarction (Nervous system disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0
Grand Mal Convlusion (Nervous system disorders) | 0 | 1
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 1 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Lobar Pneumonia (Infections and infestations) | 0 | 2
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Non-cardiac Chest Pain (General disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Radius Fracture (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=509) | Milnacipran (N=516)
Constipation (Gastrointestinal disorders) | 20 | 76
Diarrhoea (Gastrointestinal disorders) | 26 | 23
Dizziness (Nervous system disorders) | 26 | 54
Dyspepsia (Gastrointestinal disorders) | 31 | 25
Fatigue (General disorders) | 22 | 31
Headache (Nervous system disorders) | 80 | 92
Hot Flush (Vascular disorders) | 18 | 56
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 7 | 40
Hypertension (Vascular disorders) | 5 | 27
Insomnia (Psychiatric disorders) | 41 | 51
Nausea (Gastrointestinal disorders) | 106 | 189
Palpitations (Cardiac disorders) | 15 | 38
Tachycardia (Cardiac disorders) | 5 | 28
Upper Respiratory Tract Infection (Infections and infestations) | 27 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor can review results communications prior to public release & can embargo communications re: results for 90 days from time submitted to sponsor for review. PI shall not disclose sponsor's confidential info. Upon sponsor's request, PI shall delete any proprietary info & shall not include raw data in pub. On sponsor's request, PI shall delay submission for any pub while sponsor files patent apps. If trial is multi-center, PI agrees that first publication shall be a multi-center pub.